CLINICAL TRIAL: NCT01413503
Title: A Phase II Study of 131I-labeled Metaiodobenzylguanidine (MIBG) for Treatment of Patients With Metastatic or Unresectable Pheochromocytoma and Related Tumors
Brief Title: A Phase II Study of 131I- Metaiodobenzylguanidine (MIBG) for Treatment of Metastatic or Unresectable Pheochromocytoma and Related Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Paul Fitzgerald, MD, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03991
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2017-12

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Pheochromocytoma; Paraganglioma; MIBG; 131I-MIBG; Resistant; Relapsed; Treatment; UCSF; Pediatric; Adult; Oncology
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Recurrence; Neoplasms | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 131I-MIBG (Experimental): Patients received 131I-MIBG 8-12 mCi/kg (maximum 500 mCi ± 10% at investigator's discretion) diluted in 25 ml of normal saline. Patients were infused intravenously through a patient's peripheral or central line over 120 minutes
  Interventions: Radiation: 131I-MIBG

INTERVENTIONS:
Radiation: 131I-MIBG — Therapeutic 131I-MIBG will be synthesized at Nuclear Diagnostic Products (NDP; Rockaway, New Jersey) with specific activities of 9-18 Ci/mmole. The therapeutic dose: 8-12 mCi/kg (maximum 1200 mCi ± 10% at investigator's discretion) will be diluted in 25 ml of normal saline, and will be infused intravenously through a patient's peripheral or central line over 120 minutes. The patient will remain in a radiation protected isolation room until radiation emissions are ≤ 2 mr/hr at a 1 meter distance or meets institutional and state guidelines. This usually takes 4-6 days. In all cases, special shielding will be equipped in the room to minimize exposure to the outside environment and personnel will observe institutional radiation safety precautions.
  Other Names: MIBG

SUMMARY:
This is an ongoing prospective Phase II clinical trial evaluating the efficacy of 131I-MIBG for the treatment of patients with metastatic or unresectable pheochromocytoma and related tumors.

DETAILED DESCRIPTION:
1. To assess the efficacy of high-dose 131I-MIBG in the treatment of patients with malignant pheochromocytoma and related tumors, with the basis of this initial examination being the percentage of patients in CR or PR, and the percentage of patients without PD for 3 years after the initial administration on 131I-MIBG therapy.
2. To describe the response rate of malignant pheochromocytoma patients treated with high-dose 131I-MIBG.
3. To describe the toxicity of high-dose 131I-MIBG in patients with malignant pheochromocytoma.
4. To describe the overall survival and failure-free survival of malignant pheochromocytoma patients treated with high-dose 131I-MIBG.
5. To determine the utility of using the serum level of Chromogranin A as a tumor marker for patients with malignant pheochromocytoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Documentation: Histologic documentation of malignant pheochromocytoma or related tumors (paraganglioma, neuroblastoma, medullary thyroid carcinoma, carcinoid tumors), not amenable to curative surgery. Any site of origin of malignant pheochromocytoma, including but not limited to: adrenal, neck, thorax, abdominal, or pelvis is allowed.
* Prior Treatment:

  * No cytotoxic chemotherapy for at least 3 weeks prior to high-dose 131I-MIBG or concurrent with high-dose 131I-MIBG.
  * > 2 weeks since major surgery.
  * > 4 weeks since completion of prior radiation therapy, as long as measurable disease lies outside the radiation port.
  * No treatment with an investigational agent concurrent or within 30 days of high-dose 131I-MIBG.
  * Patients who have received previous chemotherapy or radiation therapy must have evidence of persistent disease on 123I-MIBG scan and elevated tumor markers or measurable CT lesions before receiving high-dose 131I-MIBG.
* Metastases Excluding Eligibility: No patients with a known significant MIBG-avid parenchymal brain metastasis; leptomeningeal metastases do not exclude eligibility. Hepatic metastases exclude eligibility if they functionally impair liver function (AST or total bilirubin ≥ 2.5 times the ULN).
* Measurable Disease Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm as measured with CT scanning. Lesions < 10 mm diameter or bone lesions in the presence of demonstrable uptake of 123I-MIBG on diagnostic scanning, plus elevated levels of tumor markers that are specific for malignant pheochromocytoma: plasma catecholamines or metanephrines, urine catecholamines or metanephrines, serum chromogranin A. Lesions whose size is considered non-measurable include the following:

  * Bone lesions (see above)
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Chylothorax
  * Lesions within the chest or abdomen that are not confirmed to be pheochromocytoma by biopsy or 123I-MIBG scanning.
* 131I-MIBG or 123I-MIBG Avidity: All patients must have 123I-MIBG or 131I-MIBG whole-body scanning prior to therapy. Metastases must be avid for the isotope such that their measured gamma radiation measures ≥ twice that of background radiation.
* Subsequent 131I-MIBG Therapies: Patients must have had pain relief or a SD or PR after a prior therapy to be eligible for another therapy. Patients with PD within 9 months of the prior therapy are excluded from receiving subsequent therapy.
* Age: ≥4 years of age.
* Life Expectancy: greater than 9 months.
* Karnofsky Performance Status: 70% or higher.
* Anticoagulation: Heparin, LMW heparin, coumadin, and other anticoagulants may be used only when platelet counts are ≥ 100,000/micronL. Platelet counts will be monitored twice weekly after 131I-MIBG therapy.
* Pregnancy & Nursing: Non-pregnant and non-nursing because the effects of high-dose 131I-MIBG on the fetus/infant are unknown.
* Second Malignancies:

  * Patients with a "currently active" second malignancy, other than non-melanoma skin cancers, are not eligible.
  * Patients are not considered to have a "currently active" second malignancy if they have been cancer-free for ≥5 years.
* Intercurrent Illness: No patients with uncontrolled intercurrent illness including but not limited to: ongoing active infections, grade 3 or 4 congestive heart failure by echocardiogram, nephrotic syndrome, serum albumin < 3, significant ascites or pleural effusion, pulmonary function testing (FVC) less than 70% of predicted for age, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Required Initial Laboratory Data (Minimum Levels):

  * Neutrophil count >/= 1,000/micronL
  * Platelet count >/= 80,000/micronL
  * AST (SGOT) ≤ 2.5 x ULN
  * Total bilirubin ≤ 2.5 x ULN
  * Creatinine ≤ 2 x ULN

Exclusion Criteria:

* 1) Pregnancy & Nursing: Non-pregnant and non-nursing because the effects of high-dose 131I-MIBG on the fetus/infant are unknown.
* 2) Second Malignancies:

  * Patients with a "currently active" second malignancy, other than non-melanoma skin cancers, are not eligible.
  * Patients are not considered to have a "currently active" second malignancy if they have been cancer-free for ≥5 years
* 3) Intercurrent Illness: No patients with uncontrolled intercurrent illness including but not limited to: ongoing active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1991-05; Primary Completion 2007-09-06 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fitzgerald, Principal Investigator — UCSF School of Medicine
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Result] Gonias S, Goldsby R, Matthay KK, Hawkins R, Price D, Huberty J, Damon L, Linker C, Sznewajs A, Shiboski S, Fitzgerald P. Phase II study of high-dose [131I]metaiodobenzylguanidine therapy for patients with metastatic pheochromocytoma and paraganglioma. J Clin Oncol. 2009 Sep 1;27(25):4162-8. doi: 10.1200/JCO.2008.21.3496. Epub 2009 Jul 27. PMID 19636009

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 131I-MIBG
Started | 50
Completed | 49
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: number of evaluable participants
Groups:
- 131I-MIBG: Patients received 131I-MIBG infused intravenously through a peripheral or central line over 120 minutes.
  Of 50 patients enrolled and treated, one patient was lost to follow-up.
Arm/Group | 131I-MIBG
Number analyzed (Participants) | 49
Age, Continuous [Mean (Full Range); unit: years] | 42.6 [10.3 to 64.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete (CR), Partial (PR), or Minor (MR) Response and Without Progressive Disease
Description: Patients with complete (CR), partial (PR), or minor (MR) response and without progressive disease 1 year from initial treatment, using RECIST RESPONSE CRITERIA for measurable soft tissue tumor: CR=No Tumor (Primary or metastatic); catacholamines, metanephrines and chromogranin A all normal. PR=Primary and all measurable sites decreased >50%; number of positive bone sites decreased by >50%; bone marrow tumor decreased by 50%. MR=No new lesions; >50% reduction of any measurable lesion (primary or metastases); <25% increase in any existing lesion.
Time Frame: After 1 year from initial treatment
Measure: Count of Participants; unit: Participants
Groups:
- 131I-MIBG: Patients received 131I-MIBG infused intravenously through a peripheral or central line over 120 minutes
Arm/Group | 131I-MIBG
Number analyzed (Participants) | 49
Participants | 28

ADVERSE EVENTS:
Description: All study records, including participant charts, IND files, and staff computers, were destroyed in a flood. Partial Adverse Event information was derived from publication-PubMed ID: 19636009
Arm/Group | 131I-MIBG
All-Cause Mortality (participants affected / at risk) | 4/49
Serious Adverse Events (participants affected / at risk) | 6/49
Other Adverse Events (participants affected / at risk) | 43/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 131I-MIBG (N=49)
Bronchiolitis obliterans organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 131I-MIBG (N=49)
Neutropenia (Blood and lymphatic system disorders) | 43
Thrombocytopenia (Blood and lymphatic system disorders) | 41
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 7
Acute hypertension (Vascular disorders) | 7
Infection (Infections and infestations) | 2
Hypogonadism (Reproductive system and breast disorders) | 4
Hyperthyroidism (Endocrine disorders) | 3

LIMITATIONS AND CAVEATS:
All study data were destroyed in a flood after study completion and prior to results posting in ClinicalTrials.gov. Partial Adverse Event information was derived from publication-PubMed ID: 19636009

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes